CLINICAL TRIAL: NCT01493024
Title: Multicenter, Prospective, Randomized, Placebo-Controlled, Double-blind Dose Escalating Study of Safety, Tolerability and Pharmacodynamics of Zirconium Silicate in Chronic Kidney Disease and Moderate Kidney Dysfunction With Mild Hyperkalemia
Brief Title: Safety & Efficacy of Zirconium Silicate in Chronic Kidney Disease or Moderate Kidney Dysfunction With Mild Hyperkalemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ZS Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ZS-002
Record Dates: First submitted 2011-12-12; First posted 2011-12-15 (Estimated); Results first posted 2018-06-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Hyperkalemia; Chronic Kidney Disease; Kidney Dysfunction
MeSH Terms: conditions — Hyperkalemia; Renal Insufficiency, Chronic | interventions — zircon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (silicified microcrystalline cellulose) randomized to mimic escalating doses of experimental drug administered three times daily (TID) with meals.
  Interventions: Drug: Placebo
- Zirconium silicate (ZS) (Experimental): Randomized escalating doses (0.3g, 3g and 10g) of ZS (fractionated, protonated, microporous zirconium silicate, an oral sorbent) administered 3 times daily (tid) with meals.
  Interventions: Drug: Zirconium silicate (ZS)

INTERVENTIONS:
Drug: Zirconium silicate (ZS) — Randomized escalating doses (0.3g, 3g and 10g) of ZS (fractionated, protonated microporous Zirconium Silicate, an oral sorbent) administered 3 times daily (tid) with meals.
  Other Names: ZS-9
  Arms: Zirconium silicate (ZS)
Drug: Placebo — Randomized to mimic escalating doses of experimental drug administered 3 times daily (tid) with meals.
  Other Names: silicified microcrystalline cellulose
  Arms: Placebo

SUMMARY:
It is hypothesized that zirconium silicate is safe and well tolerated and more effective than placebo (alternative hypothesis) in lowering serum potassium levels in subjects with serum potassium between 5 - 6.0 mmol/l versus no difference between zirconium silicate and placebo (null hypothesis). It is hypothesized that zirconium silicate even up to the top dose of 10g three times a day is well tolerated.

DETAILED DESCRIPTION:
A total of 90 subjects with moderate CKD (defined as GFR between 40- 60ml/min) and mild hyperkalemia (S-K between 5-6 mmol/l) will be enrolled in the study where, in a double-blind dose-escalating fashion (three separate cohorts), they will be randomized to receive one of the doses of ZS (0.3g, 3g and 10g) or placebo, administered 3 times (tid) daily with meals. The first cohort will have 18 subjects while both of the second and third cohorts will have 36 subjects for a total of 90 subjects.

Safety and tolerability will be assessed by an Independent Data Safety Monitoring Board (DSMB) after completion of each cohort, before escalation to the next dose level will be allowed. The next dose escalation will happen no sooner than one week after the last dose of study drug at the previous dosing level has been administered. Safety stopping rules will be specified for this study. Within the first dose level (300 mg dose), 12 subjects will be randomized to receive ZS, whereas 6 subjects will be randomized to receive placebo for a total of 18 subjects in this first cohort. In the next two cohorts (3 g and 10 g doses), 24 subjects per cohort will be randomized to receive ZS, whereas 12 subjects per cohort will be randomized to receive placebo for a total of 36 subjects in each of the second and third cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent.
* Over 18 years of age.
* GFR between 40-60 ml/min as estimated by the CKD-EPI equation. After screening two additional GFR values of between 40-60ml/min must be repeated within 24 hours before inclusion is allowed.
* S-K between 5.0 - 6.0 mmol/l (inclusive) during Study Day 0.
* Ability to have repeated blood draws or effective venous catheterization.
* Women of child bearing potential must be practicing a highly effective method of birth control.

Exclusion Criteria:

* Pseudohyperkalemia such as excessive fist clinching hemolyzed blood specimen, severe leukocytosis or thrombocytosis.
* Subjects treated with lactulose, xifaxan or other non-absorbed antibiotics for hyperammonemia within the last 7 days.
* Subjects treated with resins (such as sevelamer acetate, calcium acetate or calcium carbonate, lanthanum carbonate, Sodium polystyrene sulfonate (SPS; e.g. Kayexalate®) within the last 7 days.
* Subjects with a life expectancy of less than 3 months.
* Subjects who are HIV positive.
* Subjects who are severely physically or mentally incapacitated and who in the opinion of investigator are unable to perform the subjects' tasks associated with the protocol.
* Women who are pregnant, lactating, or planning to become pregnant.
* Subjects with Ketoacidosis/Acidemia.
* Cancer within the last 5 years (other than successfully treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or early stage prostate cancer).
* Presence of any condition which, in the opinion of the investigator, places the subject at undue risk or potentially jeopardizes the quality of the data to be generated.
* Known hypersensitivity or previous anaphylaxis to Zirconium Silicate or to components thereof.
* Subjects who have cardiac arrhythmias that require immediate treatment.
* Subjects with ECG changes associated with hyperkalemia.
* Subjects with acute kidney injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-11-30 (Actual); Primary Completion 2012-05-31 (Actual); Study Completion 2012-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Rasmussen, MD, Study Chair — ZS Pharma, Inc.
Locations (9):
- United States (9):
  - Southwest Clinical Research Institute, Tempe, Arizona
  - West Coast Clinical Trials, Costa Mesa, California
  - Riverside Clinical Research, Edgewater, Florida
  - Elite Research Institute, Inc., Miami, Florida
  - Compass Research Phase 1, LLC, Orlando, Florida
  - Lakeview Medical Research, Summerfield, Florida
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Southwest Houston Research, Ltd, Houston, Texas
  - Renal Associates, P.A., San Antonio, Texas

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Saglimbene VM, Strippoli GF. Potassium binders for chronic hyperkalaemia in people with chronic kidney disease. Cochrane Database Syst Rev. 2020 Jun 26;6(6):CD013165. doi: 10.1002/14651858.CD013165.pub2. PMID 32588430

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 9 centers in the United States from 28 November 2011 to 22 May 2012.
Pre-assignment Details: Combined Placebo Group
Groups:
- Placebo: Placebo randomized to mimic escalating doses of experimental drug administered three times daily .
- Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily: Sodium zirconium cyclosilicate 0.3 g three times daily, orally as a suspension in water
- Sodium Zirconium Cyclosilicate 3 g Three Times Daily: Sodium zirconium cyclosilicate 3 g three times daily, orally as a suspension in water
- Sodium Zirconium Cyclosilicate 10 g Three Times Daily: Sodium zirconium cyclosilicate 10 g three times daily, orally as a suspension in water
Period: Overall Study
Arm/Group | Placebo | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Sodium Zirconium Cyclosilicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Started | 30 | 12 | 24 | 24
Completed | 30 | 12 | 24 | 24
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Sodium Zirconium Cyclosilicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily | Total
Number analyzed (Participants) | 30 | 12 | 24 | 24 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.7 (11.0) | 70.3 (6.9) | 72.0 (6.3) | 72.3 (11.7) | 71.1 (9.59)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Patients' gender (Female / Male) Population: Intent-To-Treat Population
  Participants
    Female | 7 | 6 | 10 | 15 | 38
    Male | 23 | 6 | 14 | 9 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 29 | 12 | 24 | 23 | 88
  Black or African American | 1 | 0 | 0 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
Serum potassium [Mean (Standard Deviation); unit: mmol/L] — Mean of the screening time points (0 hour, 30 minutes, and 1 hour) determined by the central laboratory
  mmol/L | 5.19 (0.301) | 5.25 (0.144) | 5.11 (0.328) | 5.13 (0.378) | 5.16 (0.314)
Weight at baseline [Mean (Standard Deviation); unit: kilograms] | 95.15 (22.122) | 84.76 (18.022) | 88.96 (22.002) | 86.59 (26.311) | 89.83 (22.794)
GFR at Study Day 0 [Mean (Standard Deviation); unit: mL/min/1.73 m^2] | 45.6 (9.05) | 46.2 (4.99) | 46.8 (7.14) | 43.5 (9.01) | 45.4 (8.09)

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Exponential Rate of Change in Serum Potassium (S-K) Levels Versus Placebo During the Initial 48 Hours of Study Drug Treatment
Description: The rate of fall in S-K levels during the initial 48 hours of study drug treatment between the placebo treated subjects and the ZS treated subjects measured on a log scale
Time Frame: 24 and 48 hours post first study drug dose
Population: Intent-to-treat (ITT) population: all subjects that were randomized, received any investigational product, and had S-K levels determined at 48 hours.
Measure: Mean (Standard Error); unit: log(mmol/L/hour)
Groups:
- Placebo (Combined All Three Cohorts): Placebo randomized to mimic escalating doses of experimental drug administered three times a day (TID).
Arm/Group | Placebo (Combined All Three Cohorts) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Sodium Zirconium Cyclosilicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Number analyzed (Participants) | 30 | 12 | 24 | 24
log(mmol/L/hour)
  Day2/0 Hr ( 24 hours) | 0 (NA) — A consequence of the modeling estimate when control is the reference standard | -0.00035 (0.001166) | -0.00169 (0.000932) | -0.000143 (0.000932)
  Day 3/0 Hr (48 hours) | 0 (NA) — A consequence of the modeling estimate when control is the reference standard | -0.00045 (0.000555) | -0.00089 (0.000444) | -0.00256 (0.000444)

2. Secondary Outcome: Serum Potassium (S-K) at Individual Time Points.
Description: Serum potassium (S-K) at individual time points through Study day 3/0hour.
Time Frame: First 48 hours of study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo (Combined All Three Cohorts) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Sodium Zirconium Cyclosilicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Number analyzed (Participants) | 30 | 12 | 24 | 24
mmol/L
  Baseline | 5.14 (0.358) | 5.22 (0.264) | 5.02 (0.322) | 5.05 (0.359)
  Day 1/4Hr Post 1st Dose | 4.97 (0.564) | 5.06 (0.417) | 4.93 (0.518) | 4.80 (0.466)
  Day 1/4Hr Post 2nd Dose | 4.91 (0.465) | 5.14 (0.609) | 4.80 (0.543) | 4.68 (0.420)
  Day 1/4Hr Post 3rd Dose | 4.82 (0.558) | 4.91 (0.368) | 4.68 (0.577) | 4.50 (0.397)
  Day 2/0Hr | 4.97 (0.521) | 4.90 (0.447) | 4.66 (0.434) | 4.73 (0.463)
  Day 2/4Hr Post 1st Dose | 5.03 (0.441) | 4.97 (0.363) | 4.81 (0.601) | 4.53 (0.411)
  Day 2/4Hr Post 2nd Dose | 5.02 (0.426) | 5.04 (0.417) | 4.72 (0.604) | 4.43 (0.460)
  Day 2/4Hr Post 3rd Dose | 4.87 (0.486) | 4.83 (0.526) | 4.60 (0.566) | 4.13 (0.388)
  Day 3/0Hr | 4.94 (0.549) | 4.92 (0.506) | 4.68 (0.491) | 4.37 (0.448)
  Day 1/30 Min Post 1st Dose | 5.17 (0.419) | 5.25 (0.476) | 5.09 (0.624) | 5.03 (0.456)
  Day 1/1 Hour Post 1st Dose | 5.26 (0.524) | 5.23 (0.535) | 5.03 (0.565) | 4.94 (0.438)
  Day 1/2 Hour Post 1st Dose | 5.12 (0.532) | 5.35 (0.505) | 5.05 (0.667) | 4.93 (0.429)
  Day 2/20Hr Post 1st Dose | 4.8 (0.438) | 4.83 (0.555) | 4.60 (0.580) | 4.19 (0.378)

3. Secondary Outcome: Time Specific S-K Levels to Normalization
Description: Percent of subjects achieving S-K normalization (<=as defined by S-K levels of 3.5 to 4.9 mmol/L) from baseline at Study Days 2 and 3 at 0 hr.
Time Frame: 48 and 72 hours post first study drug dose
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Combined All Three Cohorts) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Sodium Zirconium Cyclosilicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Number analyzed (Participants) | 30 | 12 | 24 | 24
percentage of participants
  Day2/0Hr | 90 | 75 | 95.8 | 100
  Day 3/0Hr | 90 | 100 | 95.8 | 100

4. Secondary Outcome: Time Specific Decreases in S-K Levels of > = 0.5 mmol/L
Description: Percentage of participants achieving a 0.5mmol/L drop from baseline at Study Days 2 and 3 at 0 hr.
Time Frame: 24 and 48 hours post first study drug dose
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Combined All Three Cohorts) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Sodium Zirconium Cyclosilicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Number analyzed (Participants) | 30 | 12 | 24 | 24
percentage of participants
  Day 2/0Hr | 16.7 | 33.3 | 37.5 | 33.3
  Day 3/0Hr | 26.7 | 41.7 | 41.7 | 62.5

5. Secondary Outcome: Percentage of Participants With Normal S-K Levels at End of Study Day 2
Description: Percentage (%) of subjects who achieve S-K normalization at end of Study Day 2
Time Frame: 48 hours post first study drug dose
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Combined All Three Cohorts) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Sodium Zirconium Cyclosilicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Number analyzed (Participants) | 30 | 12 | 24 | 24
percentage of participants | 90 | 75 | 95.8 | 100

6. Secondary Outcome: Urine Sodium Excretion
Description: Urine sodium excretion compared between the combined placebo-treated controls and the ZS-treated subjects (measured throughout two 24-hour periods on Study Days 1 and 2).
Time Frame: 24 and 48 hours post first study drug dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo (Combined All Three Cohorts) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Sodium Zirconium Cyclosilicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Number analyzed (Participants) | 30 | 12 | 24 | 24
mmol/L
  Baseline | 91.5 (30.31) | 73.5 (29.79) | 81.7 (33.16) | 74.5 (34.20)
  Day 1/0-24Hr | 74.4 (24.8) | 66.7 (18.49) | 66.8 (26.26) | 67.1 (29.19)
  Day 2/24-48Hr | 80.1 (28.21) | 67.5 (26.63) | 71.6 (31.61) | 75.8 (35.74)

7. Secondary Outcome: Urine Potassium Excretion
Description: Urine potassium excretion compared between the combined placebo-treated controls and the ZS-treated subjects (measured throughout two 24-hour periods on Study Days 1 and 2).
Time Frame: 24 and 48 hours post study drug dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo (Combined All Three Cohorts) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Sodium Zirconium Cyclosilicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Number analyzed (Participants) | 30 | 12 | 24 | 24
mmol/L
  Baseline | 36.6 (12.47) | 32.2 (2.12) | 38.3 (11.82) | 30.3 (15.81)
  Day1/0-24Hr | 28.7 (6.41) | 32.0 (3.16) | 30.6 (5.96) | 19.7 (9.69)
  Day2/24-48Hr | 29.2 (6.42) | 31.0 (0.00) | 30.5 (6.51) | 16.9 (8.80)

8. Secondary Outcome: Urea Nitrogen Excretion
Description: Urea nitrogen excretion compared between the combined placebo-treated controls and the ZS-treated subjects (measured throughout two 24-hour periods on Study Days 1 and 2).
Time Frame: 24 and 48 hours post study drug dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo (Combined All Three Cohorts) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Sodium Zirconium Cyclosilicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Number analyzed (Participants) | 30 | 12 | 24 | 24
mg/dL
  Baseline | 525.0 (219.79) | 430.2 (162.92) | 481.0 (198.92) | 424.7 (171.88)
  Day1/ 0-24 HR | 389.2 (179.91) | 401.8 (265.74) | 414.1 (177.54) | 368.5 (147.37)
  Day2/ 24-48 HR | 460.9 (175.09) | 337.6 (115.06) | 477.0 (157.04) | 416.6 (219.56)

9. Secondary Outcome: Blood Urea Nitrogen
Description: Blood urea nitrogen compared between the combined placebo-treated controls and the ZS-treated subjects (measured 24 & 48 hours post dose on Study Days 2 and 3).
Time Frame: 24 and 48 hours post study drug dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo (Combined All Three Cohorts) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Sodium Zirconium Cyclosilicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Number analyzed (Participants) | 30 | 12 | 24 | 24
mg/dL
  Baseline | 24.50 (7.481) | 23.52 (8.217) | 25.16 (8.065) | 30.37 (8.092)
  Day 2/)0Hr | 24.05 (7.626) | 23.63 (7.241) | 23.98 (7.619) | 27.53 (7.602)
  Day 3/0Hr | 24.50 (7.284) | 23.33 (7.895) | 24.04 (7.661) | 25.60 (7.942)

10. Secondary Outcome: Serum Magnesium (S-Mg) Levels
Description: Serum magnesium compared between the combined placebo-treated controls and the ZS-treated subjects (measured at 24 & 48 hours post dose on Study Days 2 and 3).
Time Frame: 24 and 48 hours post study drug dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo (Combined All Three Cohorts) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Sodium Zirconium Cyclosilicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Number analyzed (Participants) | 30 | 12 | 24 | 24
mg/dL
  Baseline | 1.93 (0.258) | 1.95 (0.327) | 1.93 (0.143) | 1.85 (0.235)
  Day 2/0Hr | 1.92 (0.197) | 1.93 (0.271) | 1.94 (0.182) | 1.81 (0.225)
  Day 3/0Hr | 1.90 (0.204) | 1.89 (0.257) | 1.94 (0.179) | 1.83 (0.218)

11. Secondary Outcome: Serum Calcium (S-Ca) Levels
Description: Serum calcium compared between the combined placebo-treated controls and the ZS-treated subjects (measured at 24 & 48 hours post dose on Study Days 2 and 3).
Time Frame: 24 and 48 hours post study drug dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo (Combined All Three Cohorts) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Sodium Zirconium Cyclosilicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Number analyzed (Participants) | 30 | 12 | 24 | 24
mg/dL
  Baseline | 9.46 (0.595) | 9.37 (0.341) | 9.48 (0.337) | 9.50 (0.469)
  Day 2/0 Hr | 9.39 (0.439) | 9.36 (0.507) | 9.33 (0.388) | 9.22 (0.466)
  Day 3/0 hr | 9.51 (0.544) | 9.33 (0.360) | 9.30 (0.397) | 9.05 (0.425)

12. Secondary Outcome: Serum Sodium (S-Na) Levels
Description: Serum sodium compared between the combined placebo-treated controls and the ZS-treated subjects (measured at 24 & 48 hours post dose on Study Days 2 and 3).
Time Frame: 24 and 48 hours post study drug dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo (Combined All Three Cohorts) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Sodium Zirconium Cyclosilicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Number analyzed (Participants) | 30 | 12 | 24 | 24
mmol/L
  Baseline | 139.4 (2.84) | 139.1 (3.65) | 140.0 (3.09) | 137.7 (3.45)
  Day 2/0 hr | 140.1 (3.24) | 138.8 (2.04) | 140.1 (3.83) | 138.6 (3.37)
  Day 3/0 hr | 140.0 (3.36) | 138.5 (2.28) | 140.0 (3.91) | 139.6 (3.50)

13. Secondary Outcome: Serum Bicarbonate (HCO3) Levels
Description: Serum bicarbonate compared between the combined placebo-treated controls and the ZS-treated subjects (measured at 24 & 48 hours post dose on Study Days 2 and 3).
Time Frame: 24 and 48 hours post study drug dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Zirconium Silicate 3 g Three Times Daily: Zirconium Silicate (ZS) 3 g TID, three times daily as a suspension in water
Arm/Group | Placebo (Combined All Three Cohorts) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Zirconium Silicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Number analyzed (Participants) | 30 | 12 | 24 | 24
mmol/L
  Baseline | 28.1 (2.99) | 28.6 (3.11) | 28.1 (3.26) | 27.4 (3.58)
  Day 2/0 hr | 28.6 (2.46) | 29.2 (3.51) | 28.3 (3.15) | 30.1 (1.79)
  Day 3/0 hr | 29.0 (3.66) | 28.3 (2.96) | 28.7 (3.25) | 30.1 (2.31)

14. Secondary Outcome: 24-hour Urinary Excretion of Potassium
Description: 24-hour urinary excretion of potassium on Study Days 1 and Day 2
Time Frame: 24 and 48 hours post study drug dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/24 hour
Arm/Group | Placebo (Combined All Three Cohorts) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Zirconium Silicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Number analyzed (Participants) | 30 | 12 | 24 | 24
mmol/24 hour
  Baseline | 56.5 (33.96) | 62.4 (31.51) | 58.9 (20.44) | 46.9 (23.67)
  Study Day 1 | 64.7 (28.02) | 89.4 (46.62) | 60.5 (25.42) | 41.0 (20.49)
  Study Day 2 | 65.4 (29.23) | 86.6 (52.64) | 58.1 (24.77) | 31.1 (16.55)

15. Secondary Outcome: 24-hour Urinary Excretion of Sodium
Description: 24-hour urinary excretion of sodium on Study Days 1 and Day 2
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/24 hour
Arm/Group | Placebo (Combined All Three Cohorts) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Zirconium Silicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Number analyzed (Participants) | 30 | 12 | 24 | 24
mmol/24 hour
  Baseline | 145 (93.05) | 132.8 (51.09) | 124.0 (46.24) | 114.8 (49.0)
  Study Day 1 | 169.4 (88.90) | 173.7 (64.02) | 136.6 (79.5) | 141.0 (68.05)
  Study Day 2 | 181.8 (101.42) | 181.5 (101.63) | 132.5 (63.06) | 140.2 (66.86)

16. Secondary Outcome: 24-hour Urinary Excretion of Urea Nitrogen
Description: 24-hour urinary excretion of urea nitrogen on Study Days 1 and Day 2
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/24 hour
Arm/Group | Placebo (Combined All Three Cohorts) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Zirconium Silicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Number analyzed (Participants) | 30 | 12 | 24 | 24
g/24 hour
  Baseline | 7.66 (3.622) | 7.59 (2.768) | 7.03 (2.679) | 6.74 (2.618)
  Day 1 | 8.30 (3.832) | 8.51 (5.549) | 7.99 (3.929) | 7.80 (3.460)
  Day 2 | 10.37 (6.585) | 8.68 (2.475) | 8.57 (3.453) | 7.49 (3.077)

17. Secondary Outcome: 24-hour Urinary Excretion of Creatinine
Description: 24-hour urinary excretion of creatinine on Study Days 1 and Day 2
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/24 hour
Arm/Group | Placebo (Combined All Three Cohorts) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Sodium Zirconium Cyclosilicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
Number analyzed (Participants) | 30 | 12 | 24 | 24
mg/24 hour
  Baseline | 1175.39 (482.708) | 1149.00 (483.740) | 1126.26 (446.745) | 1015.67 (471.275)
  Day 1 | 1157.12 (506.515) | 1027.50 (301.315) | 996.45 (442.333) | 1008.25 (428.524)
  Day 2 | 1270.71 (544.596) | 1092.23 (411.469) | 1050.29 (344.882) | 1028.79 (430.408)

ADVERSE EVENTS:
Time Frame: Study Days 1 to 7
Arm/Group | Placebo | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily | Sodium Zirconium Cyclosilicate 3 g Three Times Daily | Sodium Zirconium Cyclosilicate 10 g Three Times Daily
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/12 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/12 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 3/30 | 1/12 | 3/24 | 8/24
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=30) | Sodium Zirconium Cyclosilicate (ZS) 0.3 g Three Times Daily (N=12) | Sodium Zirconium Cyclosilicate 3 g Three Times Daily (N=24) | Sodium Zirconium Cyclosilicate 10 g Three Times Daily (N=24)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Aspartate aminotransferae increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) — All participants that had reported adverse event of urinary tract infection had screening urinalysis (Study Day 1) that was positive for bacterial culture
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
ZS Pharma has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.